CLINICAL TRIAL: NCT06782126
Title: Self-management Support After Burns: Study Protocol for a Multicenter Stepped-wedge Hybrid Type 2 Effectiveness-implementation Study
Brief Title: A Study Protocol for the Implementation and Evaluation of a Self-management Support Program in Burns Aftercare for Burn Survivors in the Netherlands
Acronym: BET
Status: Recruiting | Type: Observational
Sponsor: Martini Hospital Groningen (Other)
Collaborators: Maasstad Hospital, Rotterdam (Unknown); Rode Kruis Ziekenhuis Beverwijk (Unknown)
Responsible Party: Sponsor
Other Study IDs: nr. 2024-033, nr 2024-048; 10070022010003 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2025-01-06; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Burns
Keywords: Burns; self-management; self-care; implementation; complex intervention
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-implementation group: Burn survivors who did not receive aftercare according to the BreeZe program
- Post-implementation group: Burn survivors who received aftercare according to the BreeZe program
  Interventions: Behavioral: BreeZe (Brandwonden en Zelfmanagement)

INTERVENTIONS:
Behavioral: BreeZe (Brandwonden en Zelfmanagement) — BreeZe is a self-management support program designed to enhance burn survivors' intrinsic motivation and self-efficacy for self-management after discharge. The intervention is based on the Self-Regulation Theory framework. Key strategies include evidence-based techniques such as goal setting and pursuit, Solution-Focused Brief Therapy, and Motivational Interviewing. The program takes a positive approach to boost motivation and self-efficacy, promoting sustainable behavior change in burn aftercare. BreeZe will be implemented through various strategies, including educating healthcare professionals on self-management, training them in communication skills (e.g., motivational interviewing), and providing materials such as a decision aid tool (self-management web) and a workbook tailored to burn survivors. Burn survivors will use the web to identify and prioritize problems, set personalized goals with their healthcare professional, and create an action plan for goal attainment.
  Groups: Post-implementation group

SUMMARY:
This study aims to evaluate a new self-management support intervention for burn survivors called BreeZe. The overall goal of BreeZe is to enhance burn survivors' self-management skills in order to integrate treatment and life goals and subsequently optimize burn survivors' quality of life and health-related outcomes. The BreeZe intervention is based on the content of the ZENN intervention, an evidence-based self-management support intervention for transplant recipient patients, which we adapted to the context of burn care. The BreeZe intervention is based on the theoretical framework of the Self-Regulation Theory. The main intervention strategies are based on evidence-based techniques, namely goal setting and pursuit, Solution-Focused Brief-Therapy, and Motivational Interviewing. In practice, this means that the intervention focuses on a positive approach in order to enhance burn survivors' intrinsic motivation and self-efficacy to encourage sustainable behaviour change regarding self-management in burns aftercare. To achieve this, we will implement BreeZe using various implementation strategies. These will include educating healthcare professionals on self-management, training them in communication skills (e.g. motivational interviewing), and providing supportive materials such as a decision aid tool (i.e., self-management web) and a workbook tailored for burn survivors.

This multicenter stepped-wedge hybrid type 2 effectiveness-implementation study aims to evaluate BreeZe's effectiveness, and to evaluate the effects of our implementation approach. The study includes a pre-implementation phase (usual care), implementation phase, and a post-implementation phase (with BreeZe), and involves the three designated burn centers in the Netherlands. The phases will be rolled out sequentially from April 2024 to November 2024, and enrollment of participants concludes in July 2025.

For evaluation, this study uses the RE-AIM evaluation framework, focusing on Reach, Effectiveness, Adoption, Implementation, and Maintenance. Our co-primary outcomes are 1) BreeZe's effectiveness in improving self-management skills in burn survivors, and 2) the effects of our implementation approach on the implementation outcomes Reach, Adoption, Implementation and Maintenance. Secondary effectiveness outcomes are self-regulation, participation, dependency, and patient-centeredness for burn survivors, and self-management support skills for healthcare professionals. Data collection for burn survivors occurs at 2 weeks, 6 months, and 12 months post-discharge, using questionnaires. Data collection for healthcare professionals occurs pre-implementation, and 3, 6 and 12 months after implementation, using questionnaires, interviews, and video observations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Admission in one of the burn centers > 24 hours and/or debridement or skin graft operation
* Proficiency of the Dutch language

Exclusion Criteria:

* Acute psychiatric illness
* Cognitive limitations
* Discharge to a different healthcare institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Emergency Management of Severe Burns (EMSB) referral criteria guide the decision to refer burn patients to a specialized burn center. Criteria for referral include: 1) total burned body surface area (TBSA) >10%, 2) >5% full-thickness burns, 3) circular burns around the neck, thorax, or extremities, 4) burns around functional areas, 5) burns with other trauma, 6) chemical burns, 7) pre-existing diseases, or 8) electrical burns. Minor burns may be managed in tertiary trauma centers or non-burn facilities, but most burn survivors are either directly admitted or transferred to a burn center. In the Netherlands, approximately 800 burn survivors are admitted to one of the three designated burn centers annually. These centers meet specific criteria for expertise, facilities, and quality of care to provide optimal treatment for burn patients.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2026-07-14 (Estimated)

PRIMARY OUTCOMES:
Self-management skills | 2 weeks, 6 months, and 12 months after discharge from burn center
  The primary outcome measure is self-management skills, assessed using the revised Partners in Health (PIH) scale. This 12-item questionnaire measures self-management behavior and knowledge, with scores on a 9-point Likert scale (higher scores indicate better self-management). Two subscales are identified in the Dutch PIH: 1) knowledge and coping, and 2) recognition and management of symptoms, adherence to treatment. Higher scores reflect better self-management skills. The PIH scale has good construct validity and reliability, with Cronbach's alpha ranging from 0.82 to 0.86. Test-retest reliability, as measured by the intraclass correlation coefficient, ranges from 0.77 to 0.818 across different language versions. While no data on responsiveness is available, the PIH consistently provides valid evidence of self-management skills in patients with chronic conditions.
Reach | 12 months post-implementation
  To determine reach, participant demographics will be compared to non-participants using the Dutch Burn Repository R3. We will compare the following characteristics: sex (m/f), age (years), total body surface area burned (%), operation (yes/no), and length of stay (days).
Adoption | 12 months post-implementation
  Adoption at staff level will be assessed by comparing the total percentage of participating healthcare professionals to the total percentage of healthcare professionals who were invited to participate, which will be quantified in percentages. Participation is defined as the completion of the three training components (i.e., e-learning, face-to-face training, follow-up training).
Implementation - Intervention fidelity | 12 months post-implementation
  To gain insight into the intervention fidelity to the core components, healthcare professionals will be asked to document in patient records when they have used certain components. A convenience sample will be taken by assessing patient records to investigate how often the core components were used, which will be described using descriptive statistics.
Implementation - implementation fidelity | 12 months post-implementation
  To gain insight in the implementation fidelity to the implementation strategies, each burn center will be asked to keep track of the completion of the implementation plan, including the staff attendance to training plan and their e-learning completion rate. Implementation fidelity will be quantified using descriptive statistics.
Maintenance (individual level) | 6 and 12 months post-implementation
  Maintenance will be assessed by the healthcare professionals' self-report of continued use using the Provider REport of Sustainment Scale (PRESS). The PRESS measure is a brief, reliable, and valid three-item measure of sustainment that is both pragmatic and useable across different evidence based practices (EBPs), provider types, and settings. The PRESS captures frontline staffs' report of their clinic, team, or agency's continued use of an EBP. It is measured on a 5-point Likert scale, with higher scores indicating better maintenance.
Maintenance (setting level) | 3 and 12 months post-implementation
  Setting-level maintenance will be assessed via the Clinical Sustainability Assessment Tool (CSAT). The CSAT is a brief and reliable instrument consisting of 35 items within seven domains to assess an institution's capacity for sustaining a clinical practice. These domains include Engaged Staff & Leadership, Engaged Stakeholders, Organizational Readiness, Workflow Integration, Implementation & Training, Monitoring & Evaluation and Outcomes & Effectiveness. Each domain includes five items that are scored on a 7-point Likert scale, where 7 indicates an individual believes their institution has that domain to a great extent. Each domain has a min-max value of 5-35, with higher scores indicating better maintenance.

SECONDARY OUTCOMES:
Self-regulation skills | 2 weeks, 6 months, and 12 months after discharge from burn center
  Self-regulation skills will be measured with the Self-Regulation Assessment (SeRA). The SeRA consists of 22 items that assess four domains of self-regulation: 1) Insight in own health condition, 2) Insight in own capabilities, 3) Trust on self and apply self-regulation, 4) Organisation of help. Answers are given on a 5-point Likert scale. Mean scores are calculated per domain, with a min-max score of 0-40. A higher score on the scale indicates a better level of self-regulation skills.
Participation | 6 and 12 months after discharge from burn center
  Participation will be measured with the Measure of Experiential Aspects of Participation (MeEAP). Participants will be asked if they participate on four different life domains: 1) employment, 2) mobility, 3) sport, and 4) exercise. The response options will be used to assess both participation in the activity (yes vs. no) and the individual's satisfaction with the level of participation
Daily activities | 2 weeks, 6 months, and 12 months after discharge from burn center
  Participants will be asked if they are capable of performing their daily activities. Daily activities will be measured with one question from the 5-level EuroQoL-5D (EQ-5D-5L). Answer options are presented on a 5-point Likert scale, with a higher score indicating better capability of performing daily activities.
Self-care | 2 weeks, 6 months, and 12 months after discharge from burn center
  Participants will be asked if they are capable of performing self-care. Self-care will be measured with one question from the 5-level EuroQoL-5D (EQ-5D-5L). Answer options are presented on a 5-point Likert scale, with a higher score indicating better capability of performing self-care.
Dependency | 2 weeks, 6 months, and 12 months after discharge from burn center
  Participants will be asked if they are dependent on other people. Dependency will be assessed with a newly formulated question. Answer options are presented on a 5-point Likert scale with a min-max value of 1-5, with a higher score indicating less dependency on other people.
Return to work or school | 6 and 12 months after discharge from burn center
  Return to work or school will be measured with the Adjusted International Consortium for Health Outcomes Measurement. Participants will be asked about their daily occupation, with the following response options: 'I work 36 hours or more per week' (1), 'I work 35 hours or less per week' (2), 'I am job searching' (3), I do not have a paid job (I go to school or am studying)' (4), I do not have a paid job (retired, volunteer, stay-at-home occupation' (5), 'I cannot work because of my burn injury' (6), 'I cannot work due to other health issues' (7). Furthermore, they will be asked if their job has been adjusted since their burn injury (e.g. physical adjustments or reduced working hours), with 'yes' or 'no' as response options. Lastly, they will be asked, if suitable, how long after their burn injury they have started working or studying again.
Patient centeredness | 6 months after discharge from burn center
  Overall experience of the received care will be assessed using the Dutch translation of the subscale 'patient-centeredness' of the American Consumer Assessment of Health Plan Survey (CAHPS). Participants will be asked if they feel listened to by their healthcare professional, if sufficient time is dedicated to their concerns, if they feel healthcare professionals take them seriously, if the healthcare professionals are able to appropriately explain things, and their level of trust in the healthcare professional's competence. Answers are measured on a 4-point Likert scale resulting in min-max values between 0-20, with higher scores indicating higher satisfaction.
Cost-effectiveness | 2 weeks, 6 months, and 12 months after discharge from burn center
  To evaluate the cost-effectiveness of the intervention, the complete 5-level EuroQol-5D questionnaire will be used to measure the effectiveness for patients compared to the control and intervention group. The EQ-5D questionnaire consists of five dimensions: mobility, self-care, daily activities, pain/discomfort and anxiety/depression. The EQ-5D L also consists the EQ visual analogue scale (VAS). Answer options are given on a 5-point Likert scale.
Self-management support skills | Before implementation, 3, 6, and 12 months post-implementation
  Self-management support skills of participating healthcare professionals will be measured with the Self-efficacy and Performance in Self-management Support (SEPSS-36). The SEPSS is a 36-item questionnaire divided over 6 subscales, using a 5-point Likert-scale. Higher mean scores (overall and for subscales) indicate a higher level of self-efficacy or performance in self-management support. Min-max values for the subscales range from 0-24, and the overall min-max value range from 0-144.
Need-supportive counselling | Before implementation, 3 and 12 months post-implementation
  Need-supportive counselling will be measured using two separate taxonomies. The first taxonomy is the Coding and Observing Need-Supportive Counselling in Chronic Care Encounters (COUNSEL-CCE). The COUNSEL-CCE consists of 44 items divided into nine scales of behavioral approaches. Response options are based on a 5-point Likert scale range from 'never observed' (0) to 'all the time observed' (4). Min-max values range from 0-24, with higher scores indicating better need-supportive counselling.
Perspectives on Adoption, Implementation, and Maintenance | 6 months post-implementation
  To explore healthcare professionals' perspectives on adoption, implementation, and maintenance, we will conduct Consolidated Framework for Implementation Research (CFIR)-informed interviews with all participating healthcare professionals. These interviews will be used to provide working hypotheses to explain the degree of adoption, to explain implementation success or failure, and to explain the degree of maintenance.
Need-supportive counselling | Before implementation, 3 and 12 months post-implementation
  The second taxonomy to assess need-supportive counselling is the Nurse-Child Interaction Taxonomy (NCIT). The NCIT consists of 16 items divided over 3 subdomains, scored on a 7-point scale, with higher scores indicating better need-supportive counselling.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Red Cross Hospital Beverwijk, Beverwijk, North Holland
  - Burn Center Martini Hospital, Groningen, Provincie Groningen
  - Maasstad Hospital Rotterdam, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Spronk I, van Uden D, van Dammen L, van Baar ME, Nieuwenhuis M, Pijpe A, Visser I, van Schie C, van Zuijlen P, Haanstra T, Lansdorp CA; Dutch Burn Care, Education & Research group. Outcomes that matter most to burn patients: A national multicentre survey study in the Netherlands. Burns. 2024 Feb;50(1):31-40. doi: 10.1016/j.burns.2023.10.018. Epub 2023 Nov 10. PMID 37985268
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Caron JG, Martin Ginis KA, Rocchi M, Sweet SN. Development of the Measure of Experiential Aspects of Participation for People With Physical Disabilities. Arch Phys Med Rehabil. 2019 Jan;100(1):67-77.e2. doi: 10.1016/j.apmr.2018.08.183. Epub 2018 Sep 27. PMID 30268805
- [Background] Petkov J, Harvey P, Battersby M. The internal consistency and construct validity of the partners in health scale: validation of a patient rated chronic condition self-management measure. Qual Life Res. 2010 Sep;19(7):1079-85. doi: 10.1007/s11136-010-9661-1. Epub 2010 May 1. PMID 20437206
- [Background] Maes S, Karoly P. Self-regulation assessment and intervention in physical health and illness: A review. Appl Psychol. 2005;54:267-299. doi:10.1111/j.1464-0597.2005.00210.x.
- [Background] Dokter J, Vloemans AF, Beerthuizen GI, van der Vlies CH, Boxma H, Breederveld R, Tuinebreijer WE, Middelkoop E, van Baar ME; Dutch Burn Repository Group. Epidemiology and trends in severe burns in the Netherlands. Burns. 2014 Nov;40(7):1406-14. doi: 10.1016/j.burns.2014.03.003. Epub 2014 Apr 2. PMID 24703338
- [Background] Arah OA, ten Asbroek AH, Delnoij DM, de Koning JS, Stam PJ, Poll AH, Vriens B, Schmidt PF, Klazinga NS. Psychometric properties of the Dutch version of the Hospital-level Consumer Assessment of Health Plans Survey instrument. Health Serv Res. 2006 Feb;41(1):284-301. doi: 10.1111/j.1475-6773.2005.00462.x. PMID 16430612
- [Background] Delnoij DM, ten Asbroek G, Arah OA, de Koning JS, Stam P, Poll A, Vriens B, Schmidt P, Klazinga NS. Made in the USA: the import of American Consumer Assessment of Health Plan Surveys (CAHPS) into the Dutch social insurance system. Eur J Public Health. 2006 Dec;16(6):652-9. doi: 10.1093/eurpub/ckl023. Epub 2006 Mar 8. PMID 16524940
- [Background] Feng YS, Kohlmann T, Janssen MF, Buchholz I. Psychometric properties of the EQ-5D-5L: a systematic review of the literature. Qual Life Res. 2021 Mar;30(3):647-673. doi: 10.1007/s11136-020-02688-y. Epub 2020 Dec 7. PMID 33284428
- [Background] Mol TI, van Bennekom CAM, Scholten EWM, Visser-Meily JMA, Beckerman H, Passier PECA, Smeets RJEM, Schiphorst Preuper HR, Post MWM. The Self-Regulation Assessment (SeRA) questionnaire: development and exploratory analyses of a new patient-reported outcome measure for rehabilitation. Disabil Rehabil. 2023 Jun;45(12):2038-2045. doi: 10.1080/09638288.2022.2080289. Epub 2022 Jun 7. PMID 35672153
- [Background] Chiu TM, Tam KT, Siu CF, Chau PW, Battersby M. Validation study of a Chinese version of Partners in Health in Hong Kong (C-PIH HK). Qual Life Res. 2017 Jan;26(1):199-203. doi: 10.1007/s11136-016-1315-5. Epub 2016 May 23. PMID 27216940
- [Background] Hudon E, Chouinard MC, Krieg C, Lambert M, Joober H, Lawn S, Smith D, Lambert S, Hudon C. The French adaptation and validation of the Partners in Health (PIH) scale among patients with chronic conditions seen in primary care. PLoS One. 2019 Oct 23;14(10):e0224191. doi: 10.1371/journal.pone.0224191. eCollection 2019. PMID 31644561
- [Background] Lenferink A, Effing T, Harvey P, Battersby M, Frith P, van Beurden W, van der Palen J, Paap MC. Construct Validity of the Dutch Version of the 12-Item Partners in Health Scale: Measuring Patient Self-Management Behaviour and Knowledge in Patients with Chronic Obstructive Pulmonary Disease. PLoS One. 2016 Aug 26;11(8):e0161595. doi: 10.1371/journal.pone.0161595. eCollection 2016. PMID 27564410